CLINICAL TRIAL: NCT00485654
Title: Racial Distribution of Heterotaxy Syndrome and Effects on Clinical Outcomes Protocol
Brief Title: Racial Distribution of Heterotaxy Syndrome
Status: Terminated | Type: Observational
Why Stopped: study was terminated because study conclusions varied.
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Director Research, Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 06-198
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2008-02

CONDITIONS: Congenital Disorders
Keywords: Heterotaxy Syndrome; Intestinal Malrotation; Functional Asplenia; Complex Cyanotic heart disease
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heterotaxy Syndrome; Volvulus Of Midgut

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Heterotaxy syndrome is a heterogeneous disease that is the result of a failure of normal right-left lateralization of the abdominal and thoracic organs during development. The major clinical manifestations include intestinal malrotation, functional asplenia and complex cyanotic heart disease.

Hypothesis: There exists a yet, un-recognized, racial distribution in heterotaxy syndrome.

DETAILED DESCRIPTION:
The exact etiology of heterotaxy is unknown, but presumed to be multifactorial. While candidate genes have been suggested, no common gene has proven responsible for this constellation of lesions. Various modes of inheritance have been described. Though there are reports of familial occurrences, no reports of racial/ethnic predominance exist. We, therefore, propose to examine the racial/ethnic distribution of heterotaxy syndrome with congenital heart disease in patients treated at this institution. In addition, the investigators will determine if race/ethnicity is a factor in clinical outcomes.

Aim 1: To determine any pattern of racial/ethnic predominance within a cohort of patients with heterotaxy syndrome with congenital heart disease.

Aim 2: To correlate race/ethnicity with disparities in morbidity and mortality in patients with heterotaxy syndrome with congenital heart disease.

This study will be a retrospective, chart review of approximately 90 - 100 medical charts, conducted on the Egleston campus of Children's Healthcare of Atlanta. Charts reviewed will cover a period between January 1, 1990 and December 31, 2005.

Data to be collected includes: DOB, diagnosis, surgical procedure, surgical outcome, survival, length of hospitalization, repeat surgical intervention, incidence of hospitalization, length of inotropic support, ventilator time, infection rate, insurance provider, list of antibiotics and zip code of residence at initial admission. In addition to the above information, data to be extracted from the medical chart of a decedent will include age at death, cause of death, laboratory data at time of death and autopsy results.

ELIGIBILITY:
Inclusion Criteria:

* All medical charts diagnosed clinically and at autopsy with heterotaxy syndrome, left atrial isomerism, right atrial isomerism or situs inversus totalis with congenital heart disease over a 16 consecutive year period at Children's Healthcare of Atlanta at Egleston.

Exclusion Criteria:

* Those who do not meet Inclusion Criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be a retrospective chart review of approximately 90 - 100 medical charts, conducted on the Egleston campus of Children's Healthcare of Atlanta. Charts reviewed will cover a period between January 1, 1990 and December 31, 2005. Data to be collected includes: DOB, diagnosis, surgical procedure, surgical outcome, survival, length of hospitalization, repeat surgical intervention, incidence of hospitalization, length of inotropic support, ventilator time, infection rate, insurance provider, list of antibiotics and zip code of residence at initial admission. In addition to the above information, data to be extracted from the medical chart of a decedent will include age at death, cause of death, laboratory data at time of death and autopsy results.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 1990-01; Primary Completion 2005-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose M Cummings, DO, Principal Investigator — Sibley Heart Center Cardiology at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States